CLINICAL TRIAL: NCT03093727
Title: Functional and Genetical Characterization of Pulmonary Langerhans Cell Histiocytosis: Diagnostic and Therapeutical Implications.
Brief Title: Characterization of Pulmonary Langerhans Cell Histiocytosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-LAN-2013-39
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Langerhans Cell Histiocytoses
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very recent studies indicate that a high percentage of HCL, about 50%, have mutations in the B-RAF oncogene. The development of ultrasensitive methodologies capable of identifying these mutations in bronchoalveolar lavage will represent a significant advance in the diagnosis and treatment of these patients. An undetermined percentage of HCL does not present mutations in B-RAF. Consequently, the deep genetic analysis, through the use of techniques of massive sequencing, can favor the identification of new alterations that contribute to the development of the disease.

We hypothesized that patients with HCL may present a different inflammatory state to healthy subjects or smokers, allowing us to identify new biomarkers.

DETAILED DESCRIPTION:
The main objective of this study is to expand the genetic and pathophysiological knowledge of this disease. For this, the following points will be developed:

* Identification of mutations in the B-RAF oncogene in Spanish patients with pulmonary LCHF.
* Development of ultrasensitive genetic analysis methods capable of identifying mutations in B-RAF in bronchoalveolar lavage (BAL) samples.
* To determine if patients with mutations in the B-RAF oncogene present distinct clinical, radiological and / or functional characteristics compared to those with absence of the mutation.
* Characterization of the inflammatory profile of patients with HPCL.

ELIGIBILITY:
Inclusion criteria

* Men and women with no age limitation
* Established histiological diagnosis of histiocytosis of langerhans cells.
* HCLP-compatible clinical-radiological picture.
* Signed informed consent

Exclusion criteria

* Non-acceptance of informed consent.
* Absence in clinical history of clinical, radiological and functional variables essential for the diagnosis of HLCP.
* Psychiatric disorder or limitation for study compression (including language, socio-cultural problem, etc.).
* Radiological findings suggestive of another chronic lung disease.
* Active respiratory infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Langerhans cell histiocytosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-09-27 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mutations in the B-RAF oncogene in Langerhans histiocytosis | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain